CLINICAL TRIAL: NCT02292446
Title: An Open-label, Multi-center, Expanded Treatment Protocol (ETP) of Ruxolitinib in Patients With Polycythemia Vera Who Are Hydroxyurea Resistant or Intolerant and for Whom no Treatment Alternatives Are Available.
Brief Title: Expanded Treatment Protocol (ETP) of Ruxolitinib in Patients With Polycythemia Vera Who Were Hydroxyurea Resistant or Intolerant and for Whom no Treatment Alternatives Was Available.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424B2001X
Record Dates: First submitted 2014-11-05; First posted 2014-11-17 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia Vera; Hematologic Diseases; Myeloproliferative Disorders; INC424; Ruxolitinib; hydroxyurea resistant; adult
MeSH Terms: conditions — Polycythemia Vera; Hematologic Diseases; Myeloproliferative Disorders | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients will receive ruxolitinib at a starting dose of 10 mg twice daily which could be titrated to most appropriate dose. Dose was not to exceed 25 mg bid nor be less than 5 mg once a day
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — supplied as 5 mg, 10 mg and 20 mg tablets to be taken orally

SUMMARY:
The purpose of this open-label, single arm, multi-center Expanded Treatment Protocol (ETP) was to provide early access to ruxolitinib and evaluate safety information in patients with polycythemia vera (PV) who were hydroxyurea (HU) resistant or intolerant and who had no other standard treatment option, nor did they qualify for another clinical study for PV

ELIGIBILITY:
Inclusion Criteria:

•Confirmed diagnosis of PV according to the 2008 World Health Organization criteria, palpable spleen, Resistant to or intolerant of hydroxyurea, ECOG performance status of 0, 1 or 2; did not have access to a comparable or satisfactory alternative treatment

Exclusion Criteria:

•Inadequate liver or renal function, Significant bacterial, fungal, parasitic, or viral infection requiring treatment, Active malignancy within the past 5 years, except treated cervical intraepithelial neoplasia, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin, with no evidence for recurrence in the past 3 years., Women who were pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (60):
- Austria (3):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Wels
- Belgium (6):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Yvoir
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
- Chile (2):
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
  - Novartis Investigative Site, Santiago
- France (17):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Le Mans, Cedex 09
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Chambéry
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Meaux
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Pringy
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villejuif
- Germany (18):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Soden
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Eisenach
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Friedrichshafen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamm
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Mutlangen
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Monterrey, Nuevo León, Mexico
- Norway (2):
  - Novartis Investigative Site, Fredrikstad
  - Novartis Investigative Site, Tromsø
- Novartis Investigative Site, Lisbon, Portugal
- Sweden (2):
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Uddevalla
- Thailand (3):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 161 patients were included in the ruxolitinib arm and 100% of the patient's received the treatment
Period: Overall Study
Arm/Group | All Patients
Started | 161
Completed | 141
Not Completed | 20
Not completed — Adverse Event | 12
Not completed — Death | 1
Not completed — Disease progression | 2
Not completed — Subject/guardian decision | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 161
Age, Customized [Number; unit: participants]
  <= 60 | 52
  >60 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 96
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 128
  Asian | 3
  Other | 30
Number of participants resistant or intolerant to hydroxyurea (HU) [Number; unit: participants] — Definition of resistant or intolerant was based on physician's evaluation
  participants
    Resistant to hydroxyurea | 60
    Intolerant to hydroxyurea | 101
Number of participants' frequency of phlebotomy in 52 weeks prior to screening [Number; unit: participants]
  1 phlebotomy | 21
  2 phlebotomies | 19
  >=3 phlebotomies | 74
  Missing | 47
Number of participants' use of prior antineoplastic therapy [Number; unit: participants] — Other prior anti-neoplastic medications included busulfan, interferon, peginterferon, pipobroman, anagrelide, momelotinib, tioguanine, mercapturine and sodium phosphate
  participants
    Prior Hydroxyurea use | 160
    Prior other anti-neoplastic medications use | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events - All Grades
Description: Summary of adverse events (all grades).
Time Frame: Baseline up to approximately 26 months
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 161
Participants
  Adverse events | 143
  Serious adverse events | 26

2. Secondary Outcome: Change From Baseline in Hematocrit Levels at All Visits
Description: Change in hematocrit levels from Baseline to each visit were measured
Time Frame: Up to approximately 26 months
Population: Number of participants qualifying for evaluation of change from baseline varied across visits
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Baseline: Hematocrit level at baseline
- Post-baseline: Post-baseline hematocrit value
- Change: Change from baseline
Arm/Group | Baseline | Post-baseline | Change
Number analyzed (Participants) | 161 | 161 | 161
percentage
  Week 4: number analyzed (Participants) | 154 | 154 | 154
  Week 4 | 45.26 (5.246) | 43.70 (5.220) | -1.55 (3.652)
  Week 8: number analyzed (Participants) | 144 | 144 | 144
  Week 8 | 45.21 (5.136) | 40.73 (4.967) | -4.48 (5.055)
  Week 12: number analyzed (Participants) | 118 | 118 | 118
  Week 12 | 45.44 (5.324) | 39.97 (5.419) | -5.47 (6.522)
  Week 16: number analyzed (Participants) | 107 | 107 | 107
  Week 16 | 45.64 (5.395) | 39.32 (5.454) | -6.32 (6.928)
  Week 20: number analyzed (Participants) | 90 | 90 | 90
  Week 20 | 45.96 (5.353) | 40.47 (5.323) | -5.49 (6.840)
  Week 24: number analyzed (Participants) | 79 | 79 | 79
  Week 24 | 45.93 (5.109) | 40.32 (4.960) | -5.62 (6.073)
  Week 36: number analyzed (Participants) | 48 | 48 | 48
  Week 36 | 45.30 (4.602) | 40.43 (4.959) | -4.86 (6.184)
  Week 48: number analyzed (Participants) | 37 | 37 | 37
  Week 48 | 45.41 (4.714) | 39.82 (4.959) | -5.59 (6.318)
  Week 60: number analyzed (Participants) | 23 | 23 | 23
  Week 60 | 46.56 (5.299) | 40.60 (5.105) | 40.60 (5.929)
  Week 72: number analyzed (Participants) | 18 | 18 | 18
  Week 72 | 47.66 (5.377) | 40.59 (4.056) | -7.07 (6.388)
  Week 84: number analyzed (Participants) | 15 | 15 | 15
  Week 84 | 48.15 (5.758) | 41.93 (5.097) | -6.23 (6.492)
  Week 96: number analyzed (Participants) | 12 | 12 | 12
  Week 96 | 50.03 (4.702) | 40.82 (4.496) | -9.21 (6.861)
  EOT: number analyzed (Participants) | 154 | 154 | 154
  EOT | 45.38 (5.202) | 39.93 (5.730) | -5.45 (5.847)

3. Secondary Outcome: Change From Baseline in Spleen Length
Description: Change in spleen length from Baseline to each visit
Time Frame: Up to approximately 26 months
Population: Number of participants qualifying for evaluation of change from baseline varied across visits
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Baseline | Post-baseline | Change
Number analyzed (Participants) | 161 | 161 | 161
cm
  Week 12: number analyzed (Participants) | 105 | 105 | 105
  Week 12 | 23.92 (14.618) | 16.83 (12.931) | -7.09 (12.770)
  Week 24: number analyzed (Participants) | 75 | 75 | 75
  Week 24 | 22.66 (14.319) | 16.26 (13.896) | -6.40 (14.101)
  Week 36: number analyzed (Participants) | 43 | 43 | 43
  Week 36 | 21.87 (13.228) | 16.70 (14.419) | -5.18 (10.929)
  Week 48: number analyzed (Participants) | 36 | 36 | 36
  Week 48 | 22.14 (13.994) | 18.76 (16.880) | -3.38 (14.438)
  Week 60: number analyzed (Participants) | 23 | 23 | 23
  Week 60 | 20.00 (13.007) | 17.35 (12.357) | -2.65 (13.753)
  Week 72: number analyzed (Participants) | 17 | 17 | 17
  Week 72 | 18.41 (13.148) | 13.47 (11.441) | -4.94 (13.840)
  Week 84: number analyzed (Participants) | 14 | 14 | 14
  Week 84 | 19.57 (14.233) | 13.36 (9.443) | -6.21 (12.135)
  Week 96: number analyzed (Participants) | 12 | 12 | 12
  Week 96 | 19.92 (14.494) | 12.33 (8.026) | -7.58 (11.237)
  End of treatment: number analyzed (Participants) | 109 | 109 | 109
  End of treatment | 3.03 (3.419) | 0.54 (1.661) | -2.49 (3.025)

4. Secondary Outcome: Change From Baseline in Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS)
Description: The MPN-SAF (Appendix 6) was a disease specific questionnaire comprised of 10 items that measures fatigue related to MPN disease and the severity of nine of the most prevalent associated symptoms including: early satiety, abdominal discomfort, inactivity, concentration, night sweats, itching, bone pain, fever and weight loss. There were three recall periods used in this questionnaire, which were 24 hours for fatigue, the past week for symptoms of early satiety, abdominal discomfort, inactivity, concentration, night sweats, itching, bone pain and fever, and the past 6 months for weight loss, Each item was scored on a scale ranging from 0 (no fatigue/absent) to 10 (As bad as you can imagine/worst imaginable). The MPN-SAF TSS was computed as the average of the observed items multiplied by 10 to achieve a 0-to-100 scale.
  The MPN-SAF TSS thus had a possible score range of 0 to 100.
Time Frame: Up to approximately 26 months
Population: Number of participants qualifying for evaluation of change from baseline varied across visits
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Baseline | Post-baseline | Change
Number analyzed (Participants) | 161 | 161 | 161
scores
  Week 12: number analyzed (Participants) | 114 | 114 | 114
  Week 12 | 23.92 (14.618) | 16.83 (12.931) | -7.09 (12.770)
  Week 24: number analyzed (Participants) | 75 | 75 | 75
  Week 24 | 22.66 (14.319) | 16.26 (13.896) | -6.40 (14.101)
  Week 36: number analyzed (Participants) | 43 | 43 | 43
  Week 36 | 21.87 (13.228) | 16.70 (14.419) | -5.18 (10.929)
  Week 48: number analyzed (Participants) | 36 | 36 | 36
  Week 48 | 22.14 (13.994) | 18.76 (16.880) | -3.38 (14.438)
  Week 60: number analyzed (Participants) | 23 | 23 | 23
  Week 60 | 20.00 (13.007) | 17.35 (12.357) | -2.65 (13.753)
  Week 72: number analyzed (Participants) | 17 | 17 | 17
  Week 72 | 18.41 (13.148) | 13.47 (11.441) | -4.94 (13.840)
  Week 84: number analyzed (Participants) | 14 | 14 | 14
  Week 84 | 19.57 (14.233) | 13.36 (9.443) | -6.21 (12.135)
  Week 96: number analyzed (Participants) | 12 | 12 | 12
  Week 96 | 19.92 (14.494) | 12.33 (8.026) | -7.58 (11.237)
  End of treatment: number analyzed (Participants) | 138 | 138 | 138
  End of treatment | 22.86 (14.225) | 18.12 (15.130) | -4.74 (13.954)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 26 months
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 1/161
Serious Adverse Events (participants affected / at risk) | 26/161
Other Adverse Events (participants affected / at risk) | 107/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=161)
Anaemia (Blood and lymphatic system disorders) | 2
Bundle branch block bilateral (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Prostatitis Escherichia coli (Infections and infestations) | 1
Accident (Injury, poisoning and procedural complications) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=161)
Anaemia (Blood and lymphatic system disorders) | 35
Thrombocytosis (Blood and lymphatic system disorders) | 11
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 12
Fatigue (General disorders) | 14
Nasopharyngitis (Infections and infestations) | 9
Weight increased (Investigations) | 13
Dizziness (Nervous system disorders) | 12
Headache (Nervous system disorders) | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 13
Hypertension (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02292446/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02292446/SAP_001.pdf